CLINICAL TRIAL: NCT05316532
Title: A Novel ECCO2R Device as a Lung Protective Measure in Hypercapnic Respiratory Failure: a Prospective Multicenter Trial
Brief Title: Novel ECCO2R Device for Hypercapnic Respiratory Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Triemli Hospital, Switzerland (Unknown); Cantonal Hospital of St. Gallen (Other); Baxter International Foundation (Unknown)
Responsible Party: Principal Investigator, Matthias Hilty, PD Dr. med. Matthias Hilty, University of Zurich
Other Study IDs: BASEC-2021-00912
Record Dates: First submitted 2021-04-21; First posted 2022-04-07 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Hypercapnic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mechanically ventilated ECCO2R group: Adult, mechanically ventilated critically ill patients with respiratory failure and incapacity to sustain lung protective ventilation
  Interventions: Device: Prismalung + treatment
- Awake spontaneously breathing ECCO2R group: Awake, spontaneously breathing critically ill patients suffering from respiratory exhaustion
  Interventions: Device: Prismalung + treatment

INTERVENTIONS:
Device: Prismalung + treatment — Low-flow extracorporeal CO2 removal with or without concurrent continuous renal replacement therapy

SUMMARY:
The objective of this study is to assess the efficacy and safety of this new Prismalung+ membrane in its intended clinical setting by demonstrating a reduction in ventilatory parameters and pulmonary energy load or the successful maintenance of spontaneous breathing, respectively, the absence of the need to initiate vv-ECMO therapy, and initial survival.

DETAILED DESCRIPTION:
Our hypotheses are that decarboxylation therapy by means of the novel Prismalung+ membrane in patients with hypercapnic respiratory failure (I) allows the reduction of tidal volume, peak airway pressure, dP and pulmonary energy load (as measured by AUC over 72 hours) as compared to baseline in mechanically ventilated patients OR is associated with successful continuation of spontaneous breathing despite respiratory exhaustion (no decision to intubate), and that these patients (II) warrant no decision to initiate vv-ECMO therapy and (III) do not experience early mortality.

The primary Objectives of the study are to test our hypotheses I to III by applying the novel Prismalung+ ECCO2R device in mechanically ventilated patients and spontaneously breathing patients experiencing hypercapnic respiratory failure in a multi-central prospective trial in three experienced intensive care units in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patient: (I) Progressive respiratory failure (pH≤7.25 and/ or PaCO2 ≥9 kPa) during mechanical ventilation (II) with an inability to maintain lung protective ventilation (VT<4 mL/kg, Ppeak <30 mbar, Driving Pressure ≤12 mbar)
* OR awake spontaneously breathing patient: Respiratory exhaustion (pH≤7.25 and/or PaCO2 ≥9 kPa)
* AND Informed Consent as documented by signature

Exclusion Criteria:

* Mechanical Ventilation group: Need for v-v ECMO
* Awake spontaneously breathing group: Need for mechanical ventilation due to inability to remain un-sedated
* Thrombocytopenia (<100G/l)
* Contraindications for Heparin therapy (history of heparin antibodies, previous history of intracranial bleeding)
* Patients under 18 years of age
* Women who are pregnant or breast feeding
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, mechanically ventilated critically ill patients with respiratory failure and incapacity to sustain lung protective ventilation or respiratory exhausting awake, spontaneously breathing critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tidal volume | At timepoint 1 (72 hours)
  Tidal volume (VT [mL/kg]) in mechanically ventilated patients or no intubation in spontaneously breathing patients
Peak Pressure | At timepoint 1 (72 hours)
  Peak Pressure (Ppeak [mbar]) in mechanically ventilated patients or no intubation in spontaneously breathing patients
Driving Pressure | At timepoint 1 (72 hours)
  Driving Pressure [mbar] in mechanically ventilated patients or no intubation in spontaneously breathing patients
VV-ECMO therapy | At timepoint 2 (28 days)
  No initiation of VV-ECMO therapy
Survival | At timepoint 2 (28 days)
  Survival

SECONDARY OUTCOMES:
Secondary endpoint - respiratory mechanics | 72 hours
  Reduction in pulmonary energy load after initiation of ECCO2R as compared to baseline in mechanically ventilated patients
Secondary endpoint - complications | 28 days
  Incidence of complications such as bleeding, thrombosis, coagulatory activation as evidences by thrombocytopenia, elevated D-Dimer levels, and plasmatic coagulatory failure.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias P Matthias, PD Dr. med., Principal Investigator — University of Zurich
Locations (1):
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided